CLINICAL TRIAL: NCT04906174
Title: Effect of Materials for Subcuticular Suture (Quill® vs. Monocryl®) on Complications After Liver Resection
Brief Title: Effect of Materials for Subcuticular Suture (Quill vs. Monocryl) on Complications After Liver Resection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0258; NCI-2021-03485 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0258 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-05-12; First posted 2021-05-28 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Liver and Intrahepatic Bile Duct Neoplasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (medical record review): Patients' medical records are reviewed retrospectively.
  Interventions: Other: Electronic Health Record Review

INTERVENTIONS:
Other: Electronic Health Record Review — Medical records are reviewed

SUMMARY:
This study investigates the effect of materials used in subcuticular suture on patients' outcomes after surgery. The prevention of surgical site wound infection is important to decrease the length of hospital stay and the post-operative risk of incisional hernia, especially in patients undergoing open hepatectomy (surgical removal of the liver). The purpose of this study is to compare the impact of the use of Quill versus Monocryl for subcuticular suture on patients' outcomes after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To investigate the impact of materials for subcuticular suture (Quill versus [vs.] Monocryl) on complications after liver resection.

OUTLINE:

Patients' medical records are reviewed retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 18 years of age undergoing liver resection at MD Anderson Cancer Center from June 1, 2020 through January 31, 2021

Exclusion Criteria:

* Patients who have a history of previous abdominal surgery will be excluded
* Pregnant women will not be included in this chart review

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing liver resection at MD Anderson Cancer Center from June 1, 2020 through January 31, 2021
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-04-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of complications after liver resection | 1 year
  The impact of materials for subcuticular suture (Quill versus Monocryl) on complications after liver resection will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Nicolas Vauthey, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org